CLINICAL TRIAL: NCT06395974
Title: Fetal Renal Artery Doppler in Patients With Preeclampsia and Its Role in Prediction of Adverse Neonatal Outcomes
Brief Title: Fetal Renal Artery Doppler in Patients With Preeclampsia
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousra M. Othman, principle investigator, Assiut University
Other Study IDs: Fetal renal a./preeclampsia
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preeclampsia
  Interventions: Other: fetal ultrasound
- control
  Interventions: Other: fetal ultrasound

INTERVENTIONS:
Other: fetal ultrasound — 2D, 3D , Doppler ultrasound

SUMMARY:
Preeclampsia is a major devastating disorder affects 2:10% of pregnancies worldwide. preeclampsia may be associated with placental insufficiency which may cause fetal blood redistribution to essential organs like brain, heart, kidney.

DETAILED DESCRIPTION:
Preeclampsia is a major devastating medical condition that affects pregnant women after 20 weeks of pregnancy. It affects 2:10% of pregnancies worldwide according to World Health Organisation with higher incidence in developing countries.

Vascular endothelial dysfunction due to abnormal placentation is believed to be the main cause of multi-organ failure and uteroplacental insufficiency that occur in preeclampsia leading to major adverse effects in both mother and fetus.

Placental insufficiency causes a redistribution of fetal blood to essential organs ; brain, heart and adrenal glands by decreasing their vascular resistance on expense of peripheral organs such as kidney which exhibit increased vascular resistance and impaired perfusion. This is in contrast to normal pregnancies near term in which renal vascular resistance falls and increased blood flow to the kidneys is observed. Doppler ultrasound examination of vasculature of selected organs such as kidneys may have a role in detection of hemodynamic rearrangements that occur in cases of placental insufficiency and preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* a) Preeclampsia:

  * Women with preeclampsia >28 weeks of pregnancy.
  * Singleton pregnancy.
  * Women with intrauterine growth restriction and abnormal amniotic fluid volume to simulate real world data.

    b) Control:
  * Women with healthy pregnancy matched by closest gestational age.

Exclusion Criteria:

* ● Multiple pregnancy.

  * Known Congenital fetal malformations.
  * Women with other comorbidity such as ischemic heart disease, DM, Autoimmune disorders, kidney disease, neurological disorders, liver or haematological disorders.
  * Women unable to provide informed consent.
  * Women who refuse to participate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: pregnant women with preeclampsia and healthy pregnant women
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
fetal renal artery doppler indices | 1 year
  the difference between the Fetal renal artery Doppler indices between preeclamptic patients and women with healthy pregnancy
Middle cerberal artery doppler indices , Umbilical artery doppler indices and placental volume | 1 year

SECONDARY OUTCOMES:
neonatal outcome | 1 year
  the ability of Fetal renal artery Doppler in prediction of neonatal complications.

CONTACTS AND LOCATIONS:
Overall Officials: Yousra O Mokhtar, Principal Investigator — principle investigator
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filipek A, Jurewicz E. [Preeclampsia - a disease of pregnant women]. Postepy Biochem. 2018 Dec 29;64(4):232-229. doi: 10.18388/pb.2018_146. Polish. PMID 30656917
- [Background] Mou AD, Barman Z, Hasan M, Miah R, Hafsa JM, Das Trisha A, Ali N. Prevalence of preeclampsia and the associated risk factors among pregnant women in Bangladesh. Sci Rep. 2021 Oct 29;11(1):21339. doi: 10.1038/s41598-021-00839-w. PMID 34716385
- [Background] Rana S, Lemoine E, Granger JP, Karumanchi SA. Preeclampsia: Pathophysiology, Challenges, and Perspectives. Circ Res. 2019 Mar 29;124(7):1094-1112. doi: 10.1161/CIRCRESAHA.118.313276. PMID 30920918
- [Background] Stigter RH, Mulder EJ, Bruinse HW, Visser GH. Doppler studies on the fetal renal artery in the severely growth-restricted fetus. Ultrasound Obstet Gynecol. 2001 Aug;18(2):141-5. doi: 10.1046/j.1469-0705.2001.00493.x. PMID 11529994
- [Background] Suranyi A, Streitman K, Pal A, Nyari T, Retz C, Foidart JM, Schaaps JP, Kovacs L. Fetal renal artery flow and renal echogenicity in the chronically hypoxic state. Pediatr Nephrol. 2000 May;14(5):393-9. doi: 10.1007/s004670050781. PMID 10805467
- [Background] Nicolaides K, Giuseppe R, Hecher K, Ximenes R. Doppler in Obstetrics. ISUOG Educational Series, The Fetal Medicine Foundation, 2022.
- [Background] Ma'ayeh M, Krishnan V, Gee SE, Russo J, Shellhaas C, Rood KM. Fetal renal artery impedance in pregnancies affected by preeclampsia. J Perinat Med. 2020 Mar 14:/j/jpme.ahead-of-print/jpm-2020-0024/jpm-2020-0024.xml. doi: 10.1515/jpm-2020-0024. Online ahead of print. PMID 32171001
- [Background] Gestational Hypertension and Preeclampsia: ACOG Practice Bulletin, Number 222. Obstet Gynecol. 2020 Jun;135(6):e237-e260. doi: 10.1097/AOG.0000000000003891. PMID 32443079
- [Background] Azpurua H, Dulay AT, Buhimschi IA, Bahtiyar MO, Funai E, Abdel-Razeq SS, Luo G, Bhandari V, Copel JA, Buhimschi CS. Fetal renal artery impedance as assessed by Doppler ultrasound in pregnancies complicated by intraamniotic inflammation and preterm birth. Am J Obstet Gynecol. 2009 Feb;200(2):203.e1-11. doi: 10.1016/j.ajog.2008.11.001. PMID 19185102
- [Background] Magee LA, Nicolaides KH, von Dadelszen P. Preeclampsia. N Engl J Med. 2022 May 12;386(19):1817-1832. doi: 10.1056/NEJMra2109523. No abstract available. PMID 35544388